CLINICAL TRIAL: NCT05544331
Title: Comparison of Written and Video Home Exercise Program in the Patients With Chronic Symptomatic Lumbar Disc Herniation
Brief Title: Rehabilitation in Lumbar Disc Herniation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tugce Ozen, research assistant, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2021.351
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Symptomatic Lumbar Disc Herniation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Written exercise group (Experimental): The exercise program will consist of core stabilization exercises, which target various trunk muscles to optimize segmental control, spinal stability, spinal stiffness, orientation and the interoperability of these features. The exercise program will be in writing form, which is a common home exercise program type.
  Interventions: Behavioral: Exercise group (written form)
- Video based exercise group (Experimental): The exercise program will consist of core stabilization exercises, which provide segmental control optimization, spinal stabilization, spinal stiffness, orientation and the interoperability of these features. The exercise program will be given patients as video records, which provide visual and auditory feedbacks.
  Interventions: Behavioral: Exercise group (video based)
- Control group (No Intervention): The patients, who are referred and will wait for the exercise program in their routine daily life. Measurements will be performed at the same time frame in experimental group. After the 12 weeks of follow up period, they will join the exercise program.

INTERVENTIONS:
Behavioral: Exercise group (written form) — The exercise program will be structUred with core stabilization exercises. Patients will be given the written form of exercises and will be applied as home exercises. Exercise progression will be provided by position changes.
  Arms: Written exercise group
Behavioral: Exercise group (video based) — The exercise program will be structUred with core stabilization exercises. Patients will be given the exercise videos, which provide visual and auditory feedback, and will be applied as home exercises. Exercise progression will be provided by position changes.
  Arms: Video based exercise group

SUMMARY:
The aim of this study is to compare the effects of written and video based home exercise program in patients with symptomatic lumbar disc herniation on pain level, function and quality of life.

DETAILED DESCRIPTION:
45 symptomatic lumbar disc herniation patients, who are in chronic period and aged between 18-65 years, will be included. The participants will be randomised into three groups. 15 patients will be included in the written home exercise group,15 patients will be in video based home exercise group and 15 patients in the control group. In the written exercise group and video based exercise group, exercise programs will be 8 weeks. In the control group, the exercise protocol will not be performed during 8 weeks.

The outcomes will include the quality of life, pain level, functional capacity, kinesiophobia. In the exercise groups, the evaluations will be made in the first interview (before exercise program), at the end of 8 weeks of exercise (when the exercise program is completed) and in 12th weeks (4 weeks after the exercise program completion). Evaluations in the control group will be carried out at the first interview, at the 8th week, 12th weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged between of 18-65 years
* Having been diagnosed with a lumbar disc herniation
* No need for surgery due to lumbar disc herniation
* Having pain in the lower back or leg for at least 12 weeks
* Not using corticosteroids
* To be oriented and cooperative
* To be volunteer to participate in the study

Exclusion Criteria:

* Having undergone lumbar spine surgery
* Having undergone lower extremity, upper extremity, spine surgery in the last 1 year
* Presence of lumbar stenosis
* Analgesic addiction, or any addiction
* Presence of tumor
* Presence of metastases
* Presence of rheumatological diseases
* The presence of scoliosis, congenital deformity
* Presence of leg length discrepancy
* Being pregnant
* To have uncontrolled hypertension
* To have exercise-dependent angina

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Disability | Change from baseline at week 8, and 12.week.
  Oswestry Disability Index (ODI) will be used to evaluate patients perceptions of low back related disability. ODI consists of 10 questions, scored between 0 and 5.
Pain perception | Change from baseline at week 8, and12.week.
  Numeric Rated Scale (NRS) will be used to evaluate pain perception. Patients will be asked rated their pain between 0 and 10.
Kinesiophobia | Change from baseline at week 8, and12.week.
  Tampa Kinesiophobia Scale will be used. It consists of 17 questions about fear of movement and reinjury. Each question scored between 1 and 4.
Emotional status | Change from baseline at week 8, and12.week.
  Hospital Anxiety and Depression Scale (HADS) will be used for evaluate the patients' anxiety and depression status. HADS consists of 14 questions, which scored between 1 and 3.
Health related quality of life | Change from baseline at week 8, and12.week.
  SF-36 Health Related Quality of Life (SF-36) questionnaire will be used. SF-36 consists of 36 questions and evaluate different aspects of quality of life.
Range of motion of lumbar spine | Change from baseline at week 8, and12.week.
  The range of lumbar flexion and extension will be measured by the inclinometer. While the person is standing on both feet, first the inclinometer will be placed on the reference points on the spine. For lumbar flexion value The person will be asked to bend forward as much as he can without bending his legs. For extension value, the person will be asked to bend backwards as much as possible without bending his legs, and at the last point, the inclinometer will be read and the value will be recorded.
  Lumbar lordosis will be measured by the inclinometer. While the patients stands with his feet shoulder-width apart and knees straight, the measurement will be taken by the inclinometer placed on the reference points.
Flexibility | Change from baseline at week 8, and12.week.
  Fingertip-to-Floor Test will be applied. The person will be asked to lean forward without bending their knees while standing on a high platform, and the distance between the fingertip and the platform will be measured. Values will be recorded as centimeter.
  Side bending test will be used to measure the flexibility of spine in right and left lateral flexion. The patient will be asked to bend his back to the right and left sides, without separating his back from the wall. The results will be recorded as centimeter.
Static endurance | Change from baseline at week 8, and12.week.
  Lateral Bridge Test will be used to evaluate the static endurance of the lateral core muscles. The subjects will be asked to turn on their right side, raise their body on their forearms and toes and keep them in this position, and the time until the position deteriorates will be recorded as second.
  Sorensen Test will be used to evaluate the static endurance of trunk extensors. The subjects were positioned in the prone position, with the pelvis, hips and knees on the bed. The subjects will be asked to extend their upper body straight forward from the edge of the table and the time until the deterioration of the straight position is recorded.
  Trunk Flexors Endurance Test will be used to evaluate static endurance of the trunk flexors. The subjects were positioned with the trunk in 60 degree flexion, knees and hips in 90 degree flexion position.When the 60 degree trunk flexion is impaired, the test will be terminated and the time will be recorded.
Dynamic endurance | Change from baseline at week 8, and12.week.
  Sit-ups' Test will be used to evaluate the endurance of the abdominal muscles. The patients will be asked to flex the trunk while the knees are in the flexed position and the feet are stabilized. Each test of the patients is 30 seconds. The number of times they can do it will be recorded.
  Modified 'Push-ups' Test will be used to evaluate the upper body strength endurance. Subjects will be asked to lift the head, shoulders and trunk from the ground in the prone position with the arms and elbows flexed and the elbows fully extended. During the test, the knees will be positioned in flexion (25). Each test of the patients is 30 seconds. The number of times they can do it will be recorded.
Exercise adherence | Change from baseline at week 8, and12.week.
  The patients will be asked to note the number of the days they exercise in each week.

CONTACTS AND LOCATIONS:
Overall Officials: Tugce Ozen, MSc, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)